CLINICAL TRIAL: NCT06403449
Title: The Effectiveness of Group-Delivered Guided Written Exposure Therapy for PTSD and Subclinical PTSD Among Chinese Adolescents: a Pilot Randomized Controlled Trial
Brief Title: The Effectiveness of Group-Delivered Guided Written Exposure Therapy for PTSD and Subclinical PTSD Among Adolescents : a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Research Fellow, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-WET on Adolescents PTSD
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-05

CONDITIONS: PTSD
Keywords: PTSD; adolescents; randomized controlled trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Waiting Lists

STUDY DESIGN:
Masking Description: Randomization was conducted by an independent research assistant, and the random sequence was concealed from the investigator until the process was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G-WET (Experimental)
  Interventions: Behavioral: Group-delivered guided written exposure therapy-revised version
- Waiting-List (WL) condition (Other)
  Interventions: Behavioral: Waiting-List (WL) condition

INTERVENTIONS:
Behavioral: Group-delivered guided written exposure therapy-revised version — Group-Delivered guided WET-R (G-WET) is a manualized exposure-based therapy program consisting of 5-8 sequential sessions. The interval between every 2 consecutive sessions is 0-2 days. There will be 5-8 group-delivered sessions in total (only one index trauma will be discussed), and 1-2 weeks to complete.The first and last sessions are scheduled to last for 1.5 hours each, while the other sessions will be 50 minutes in duration.
  Arms: G-WET
Behavioral: Waiting-List (WL) condition — Participants assigned to WL will be asked to not work with other therapists or seek additional treatment for trauma-related difficulties during the 2-week WL period. After the one-month follow-up of the WET-R group, they will receive the same treatment (Group-Delivered guided written exposure therapy-revised version).WL participants will also be given contact information to use in case of worsening symptoms or increasing distress.
  Arms: Waiting-List (WL) condition

SUMMARY:
The study aims to examine the effectiveness of the group-delivered guided written exposure therapy (G-WET) for post-traumatic stress disorder (PTSD) and subclinical PTSD among Chinese adolescents with a randomized controlled trial. The study will recruit 40 participants, with 20 randomized to the G-WET group and 20 randomized to the waiting list (WL) group. The G-WET intervention consists of 5-8 group sessions. The primary outcome PCL-5 ( PTSD Checklist-5) will be administered on baseline, post-treatment, 1-month follow-up, 3-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 10-18 years.
2. Meeting full or subthreshold PTSD (up to one symptom missing) diagnostic criteria according to the Child PTSD Symptom Scale-Interview Version for DSM-5 (CPSS-5-I).
3. If taking psychotropic medication, currently stabilized on psychotropic medication for at least four weeks.
4. Capable of writing and understanding written instructions.

Exclusion Criteria:

1. Presence of severe psychopathology necessitating immediate medical attention
2. Moderate to high suicide risk (e.g., intent or plan to attempt suicide in the near future)
3. Evidence of a moderate or severe traumatic brain injury
4. Currently undergoing psychotherapy specifically for PTSD.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist-5 (PCL-5) | baseline, post treatment(2 weeks), 6 weeks, 14 weeks
  PCL-5 was a 20-item self-report scale that assesses PTSD DSM-5 diagnosis and symptom severity in the past month. Items were rated on a 5-point Likert scale from 0 ("not at all") to 4("extremely").The Chinese version of PCL-5 has shown good psychometric properties in trauma-affected Chinese adolescents.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9-item | baseline, post treatment(2 weeks), 6 weeks, 14 weeks
  Patient Health Questionnaire 9-item (PHQ-9), a self-report measure for depressive symptoms in past two weeks, comprises 9 items rated from 0 (not at all) to 3 (nearly every day). The PHQ-9 has good psychometric properties in Chinese adolescents.
Generalized Anxiety Disorder 7-item | baseline, post treatment(2 weeks), 6 weeks, 14 weeks
  Generalized Anxiety Disorder 7-item (GAD-7) scale is a 7- item self-report measure assess anxiety symptoms in past two weeks. Each item is rated from 0 (not at all) to 3 (nearly every day).The Chinese version GAD-7 score has good psychometric properties among adolescents.
The Strengths and Difficulties Questionnaire | baseline, post treatment(2 weeks), 6 weeks, 14 weeks
  The Strengths and Difficulties Questionnaire (SDQ) is a 25-item self-report questionnaire assessing emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviour .The response scale ranges from 0 ( not true) to 2 (certainly true). Chinese version has been demonstrated to have good internal consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided